CLINICAL TRIAL: NCT01110291
Title: Activity of CYP3A and Genotypes of CYP3A5 and MDR1 as Predictors of the Clearance and Adverse Effects of Docetaxel, and the Effect of Docetaxel to CYP3A Activity in Previously Untreated Breast Cancer Patients
Brief Title: Study of Usefulness of Genotyping to Predict Docetaxel Exposure and Adverse Events
Acronym: Docetaxel
Status: Completed | Type: Observational
Sponsor: University of Turku (Other)
Collaborators: Sanofi (Industry); Turku University Hospital (Other Government); Vaasa Central Hospital, Vaasa, Finland (Other); medbase Oy Ltd (Unknown)
Responsible Party: Johanna Hilli, Department of Pharmacology, Drug Development and Therapeutics, University of Turku, Turku, Finland
Other Study IDs: XRP 6976A/6022
Record Dates: First submitted 2010-04-22; First posted 2010-04-26 (Estimated); Last update posted 2010-04-27 (Estimated); Status verified 2010-04

CONDITIONS: CYP3A Phenotyping; CYP3A5 and MDR1 Genotyping; Docetaxel Toxicity; Associations Between Genetic Data and Docetaxel Toxicity
Keywords: docetaxel toxicity; CYP3A activity; CYP3A5; MDR1; peroral midazolam
MeSH Terms: interventions — Docetaxel; CEF regimen

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples for genotyping and phenotyping as well as analysis of docetaxel concentrations.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Breast cancer: Twenty patients with verified high risk breast cancer will be included in the study.
  Interventions: Drug: docetaxel + CEF

INTERVENTIONS:
Drug: docetaxel + CEF — Docetaxel 80 mg/m² of body surface area (BSA) will be given as an i.v. infusion during 60 minutes on day 0 in a 20-day schedule. The cycle is repeated three times.
  Three weeks after the last docetaxel regimen, all patients will receive the CEF-combination treatment. In CEF-combination cyclophosphamide will be given 600 mg/m²of BSA as an i.v. infusion during 15 - 30 minutes on day 0 in a 20-day schedule. This is followed by fluorouracil given 600 mg/m² of BSA as an i.v. infusion during 15 - 30 minutes . Epirubicin will be given 60 mg/m² of BSA as an i.v. infusion during 15 - 30 minutes. This combination therapy will be repeated three times.

SUMMARY:
Twenty patients with verified high risk breast cancer will be included in the study. Patients will receive three cycles of docetaxel followed by three cycles of CEF for their adjuvant treatment. The phenotype of CYP3A and the genotype of CYP3A5 and MDR1 will be assessed. Also the effect of docetaxel in the activity of CYP3A will be measured by peroral midazolam.

Primary Object:

The primary object of this study is to define, if it is possible to predict the clearance and/ or toxicity of docetaxel by assessing

* activity of CYP3A4 by midazolam test (CYP3A4 phenotype)
* CYP3A5 genotype
* MDR1 genotype

Secondary object:

The secondary object of this study is to define whether the treatment with docetaxel alters the activity of CYP3A4 enzyme in previously untreated breast cancer patients.

ELIGIBILITY:
Inclusion Criteria:

Subjects may be included in the study only if they meet all of the following criteria:

1. The patient has received information on the purpose of the study and the meaning of the treatment, and has given verbal and written consent to participate in the study. The patient is accessible for treatment and follow-up.
2. Histologically verified diagnosis of breast cancer
3. High risk for recurrence ( node positive or node negative if T2 with histological grade 2 or 3, or Pgr negative)
4. No metastases
5. Females, age =<60
6. No concomitant regular medication which is either substrate, inducer or inhibitor of CYP3A4

Exclusion Criteria:

Subjects will be excluded from the study for any of the following reasons:

1. Poor performance status,>=2 according to WHO
2. Inadequate bone marrow reserve defined as:

   * hemoglobin < 100 g/L
   * leukocytes < 3.0 x 10E9/L or neutrophiles < 1.5 x 10E9/L
   * plateless < 120 x 10E9/L
3. Inadequate liver function defined as:

   * ALAT is > 1.5 x units of normal level
   * elevated bilirubin (unless verified Gilbert´s syndrome)
   * alkaline phosphatase is > 2.5 x units of normal level
4. History of concomitant serious physical or psychiatric disease, which makes a regular cytotoxic treatment impossible
5. cardiac insufficience; severe arrhythmia; severe hypertension; cardiac infarction within one year or other active cardiac disease
6. pregnant or lactating patients
7. abuse of alcohol or any narcotic substances

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Twenty patients with verified high risk breast cancer.
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2003-04; Primary Completion 2004-01 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
docetaxel toxicity
  There were no specific outcome measures in this study. The chemotherapy was given in a predetermined schedule and additionally blood samples were drawn for genotyping. The adverse events were recorded and compared with the data from genotyping.

SECONDARY OUTCOMES:
survival
  No specific outcome measures. Survival data was collected and compared with the data from genotyping.

CONTACTS AND LOCATIONS:
Overall Officials: Johanna Hilli, MD, PhD, Principal Investigator — Department of Pharmacology, Drug Development and Therapeutics, University of Turku, Turku, Finland; Liisa Sailas, MD, Study Chair — Department of Oncology, Vaasa Central Hospital, Vaasa, Finland; Sirkku Jyrkkiö, MD, PhD, Study Chair — Department of Oncology and Radiotherapy, Turku University Hospital, Turku, Finland; Seppo Pyrhönen, MD, PhD, Study Chair — Department of Oncology and Radiotherapy, Turku University Hospital, Turku, Finland; Kari Laine, MD, PhD, Study Chair — medbase Oy Ltd, Turku, Finland
Locations (1):
- Turku University Hospital, Turku, Finland

REFERENCES:
- [Derived] Hilli J, Sailas L, Jyrkkio S, Pyrhonen S, Laine K. NCT01110291: induction of CYP3A activity and lowered exposure to docetaxel in patients with primary breast cancer. Cancer Chemother Pharmacol. 2011 Jun;67(6):1353-62. doi: 10.1007/s00280-010-1426-6. Epub 2010 Aug 27. PMID 20798939